CLINICAL TRIAL: NCT04298073
Title: Effect of Skipping Maintenance BCG on the Recurrence and Progression of T1a Urinary Bladder Tumor.
Brief Title: Skipping BCG for T1a Urinary Bladder Tumor.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ali Hamed, dr Ahmed ali, Assiut University
Other Study IDs: new treatment bladder cancer
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Superficial Bladder Cancer t1a

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bladder cancer is the most common malignancy involving theurinary system and the ninth most common malignancy worldwide .In Egypt, the urinary bladder cancer accounted for about 31% of the total incidence of cancers that subsequently decreased to 12% in the recent years .Transitional cell (Urothelial) carcinoma is the most common type of bladder cancer, about more than 90% all bladder cancers . Other pathological types are less common such as squamous cell carcinoma (observed in about 5% of bladder cancers), adenocarcinoma (observed in approximately 1% of bladder cancers) and small cell carcinoma. Urothelial carcinomas are divided clinically into superficial tumors and muscle invasive tumors. Grossly they may appear in various forms, most commonly papillary, but may also appear as a nodule or an irregular solid growth .Accurate prediction of progression is essential need in T1 bladder cancer (BCa) because the stakes are high for this disease. About one-third of patients never recur after initial treatment, one-third have cancer that recurs as non-muscle invasive BCa (NMIBC), and one-third progress to muscle-invasive BCa with significantly worse clinical outcome . Recurrence and progression rates for pT1 tumors are highly variable Accurate prediction of progression is essential need in T1 bladder cancer management. There is difficulty in predication of T1 progression due to intrinsic difficulty in assessing the presence and extent of invasion. Patient prognosis and management have been affected by the Identification of the muscularis mucosa (MM) by Dixon and Gosling in 1983 . Elderly patients with bladder cancer frequently have comorbid conditions that make conservative management preferable for early invasive urothelial carcinomas. Several studies have explored the utility of evaluating the spatial relationship of invasive tumor to the Muscularis mucosa for sub classification of pT1 urothelial carcinomas . Muscularis mucosa consists of thin and wavy fascicles of smooth muscle frequently associated with large, thin-walled blood vessels in the submucosa of the bladder wall . It can be identified in 15-83% of biopsy specimens . T1 bladder staging has been changing and led to its classification into two groups: T1a (minimally invasive) tumors (i.e., tumors that extend into the lamina propria but are located above the level of the MM), and T1b (invasive) tumors (i.e., tumors that invade beyond the MM). Treatments for T1 bladder cancers are grouped into three categories. First, the tumour can be resected (TURBT) at the initial or restaging setting, which can be performed with white or blue-light cystoscopy. The second approach involves intravesical BCG administration with multiple years of maintenance therapy. Finally, aggressive or high risk T1 bladder cancers can be managed by radical cystectomy at 'early' or 'delayed' time points relative to diagnosis .

DETAILED DESCRIPTION:
Bladder cancer is the most common malignancy involving theurinary system and the ninth most common malignancy worldwide .In Egypt, the urinary bladder cancer accounted for about 31% of the total incidence of cancers that subsequently decreased to 12% in the recent years .Transitional cell (Urothelial) carcinoma is the most common type of bladder cancer, about more than 90% all bladder cancers . Other pathological types are less common such as squamous cell carcinoma (observed in about 5% of bladder cancers), adenocarcinoma (observed in approximately 1% of bladder cancers) and small cell carcinoma. Urothelial carcinomas are divided clinically into superficial tumors and muscle invasive tumors. Grossly they may appear in various forms, most commonly papillary, but may also appear as a nodule or an irregular solid growth .Accurate prediction of progression is essential need in T1 bladder cancer (BCa) because the stakes are high for this disease. About one-third of patients never recur after initial treatment, one-third have cancer that recurs as non-muscle invasive BCa (NMIBC), and one-third progress to muscle-invasive BCa with significantly worse clinical outcome . Recurrence and progression rates for pT1 tumors are highly variable Accurate prediction of progression is essential need in T1 bladder cancer management. There is difficulty in predication of T1 progression due to intrinsic difficulty in assessing the presence and extent of invasion. Patient prognosis and management have been affected by the Identification of the muscularis mucosa (MM) by Dixon and Gosling in 1983 . Elderly patients with bladder cancer frequently have comorbid conditions that make conservative management preferable for early invasive urothelial carcinomas. Several studies have explored the utility of evaluating the spatial relationship of invasive tumor to the Muscularis mucosa for sub classification of pT1 urothelial carcinomas . Muscularis mucosa consists of thin and wavy fascicles of smooth muscle frequently associated with large, thin-walled blood vessels in the submucosa of the bladder wall . It can be identified in 15-83% of biopsy specimens . T1 bladder staging has been changing and led to its classification into two groups: T1a (minimally invasive) tumors (i.e., tumors that extend into the lamina propria but are located above the level of the MM), and T1b (invasive) tumors (i.e., tumors that invade beyond the MM). Treatments for T1 bladder cancers are grouped into three categories. First, the tumour can be resected (TURBT) at the initial or restaging setting, which can be performed with white or blue-light cystoscopy. The second approach involves intravesical BCG administration with multiple years of maintenance therapy. Finally, aggressive or high risk T1 bladder cancers can be managed by radical cystectomy at 'early' or 'delayed' time points relative to diagnosis .

ELIGIBILITY:
Inclusion Criteria:

* The study will include all patients that diagnosed for the first time as T1a urothelial carcinoma .

Exclusion Criteria:

1. Other variants of bladder cancer as squamous cell carcinoma of urinary bladder ,small cell carcinoma of urinary bladder, -sarcomatoid variant of urinary bladder & anaplastic cell carcinoma of urinary bladder
2. patients Who were previously treated for bladder cancer by any modality including TURT, BCG, chemotherapy and radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients who attending our oncological urology outpatient clinic consented to participate in the study.
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2020-03-04 (Estimated); Primary Completion 2022-03-04 (Estimated); Study Completion 2022-04-04 (Estimated)

PRIMARY OUTCOMES:
follow up | 3 months
  evaluation if there is recurrence or progression of T1a bladder tumor.